CLINICAL TRIAL: NCT04659824
Title: Study of Iron Accumulation Measured in MRI in Non-pathological Aging
Acronym: FER-IRM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_24; 2020-A00491-38 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy

SUMMARY:
To study the correlation between the iron load in brain, measured in MRI, and the age of healthy subjects Secondary objectives are to study the correlations between the iron load in cortical brain regions and (i) the cognitive performances, (ii) markers of aging (MRI, EEG, OCT, biology),and (iii) demographical factors involved in iron load.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 95 years old
* French speaker with capability to understand the instructions
* Health insurance

Exclusion Criteria:

* Pregnancy
* minor subject
* no informed consent agreement
* subject enrolled in pharmaceutic study or exclusion period
* MRI contra-indications
* Neurological or psychiatric disorders
* MOCA < 26
* Psychotropic drugs
* More than 3 MRI exams
* More than 1 neuropsychological assessment (same cognitive tests) in the last 12 months
* Unable to follow the entire protocol according to the investigator

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects from 18 to 95 years old stratified by sex and age groups
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between iron load in MRI and age | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Grégory KUCHCINSKI, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France